CLINICAL TRIAL: NCT04022668
Title: Diagnostic Accuracy of Electrocardiogram for Acute Coronary Occlusion
Brief Title: Diagnostic Accuracy of Electrocardiogram for Acute Coronary Occlusion Resulting in Myocardial Infarction
Acronym: DIFOCCULT
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Collaborators: Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: YeditepeU001
Record Dates: First submitted 2019-07-08; First posted 2019-07-17 (Actual); Results first posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Myocardial Infarction; Acute Coronary Syndrome; Coronary Artery Disease
Keywords: Acute Coronary Occlusion; Occlusive Myocardial Infarction; Non-occlusive Myocardial Infarction; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Coronary Occlusion; Coronary Thrombosis; Myocardial Ischemia; Coronary Disease
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome; Coronary Artery Disease; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Coronary Occlusion; Coronary Thrombosis; Myocardial Ischemia; Coronary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- STEMI: Current international ECG criteria (New ST-segment elevation at the J-point in two contiguous leads with the cut-points: ≥0.1 mV millivolts (mV) in all leads other than leads V2-V3; for leads V2-V3: ≥2 mm in men ≥40 years; ≥2.5 mm in men <40 years, or ≥1.5 mm in women regardless of age) with troponin rise above 99th percentile in a clinical situation suggestive of myocardial ischemia.
  Interventions: Radiation: Coronary angiogram
- NSTEMI: Troponin rise above 99th percentile in a clinical situation suggestive of myocardial ischemia without abovementioned criteria.
  Interventions: Radiation: Coronary angiogram
- Normal: Emergency department admission with a clinical picture compatible with acute coronary syndrome, but no change in serial ECGs and no rise in cardiac biomarkers

INTERVENTIONS:
Radiation: Coronary angiogram — Routine coronary angiogram, if indicated
  Groups: NSTEMI; STEMI

SUMMARY:
The decision of emergency reperfusion of a suspected acute coronary artery occlusion by means of percutaneous coronary intervention or intravenous thrombolytics depends on the presence of a certain amount of ST-segment elevation in the electrocardiogram (ECG) as recommended by international guidelines. However, recommended ST-segment elevation cut-off values for acute coronary occlusion diagnosis are highly insensitive, and their evidence base is weak. The objective of this study is to test the accuracy of various electrocardiographic patterns (including, but not limited to, ST-segment elevation) for the diagnosis of acute coronary occlusion. This information can serve to offer an accuracy profile for various ECG findings and enable clinicians to define the ECG probability of an acute coronary occlusion according to these ECG findings and clinical picture, which in turn would provide a significant improvement in the care for patients who present to the hospital with possible coronary occlusion. The primary analysis will be designed as a single-center, retrospective case-control study.

DETAILED DESCRIPTION:
In this retrospective, single-center, case-control study the investigators will seek to compare the diagnostic accuracy of various ECG criteria to identify acute coronary occlusion (ACO). The investigators will scan the charts of the patients presenting to emergency department with a clinical picture suggestive of acute coronary syndrome in the specified time period. Patients without any admission ECG will be excluded. Patients who had a final diagnosis of myocardial infarction (MI) with or without subsequent coronary intervention will be enrolled. These patients will be classified as ST-segment elevation (STEMI) group or non-ST-segment elevation (NSTEMI) group according to their final diagnosis. Patient who had been excluded for acute coronary syndrome with serial unchanging ECGs AND negative serial troponins will constitute a third group. Allocation to each group will be continued until the patient number in each group reaches up to 1000 patients. The dead or alive status of all included patients will be checked from the electronic national database.

All ECGs will be reviewed by two cardiologists blinded to the angiographic and clinical outcomes. The presence of predefined ECG findings of ACO (including, but not limited to, current established STEMI criteria) will be recorded. The coronary angiograms of the first two groups will be reviewed for ACO by independent investigators who are blinded to ECG parameters. The diagnosis of acute coronary occlusion will be dependent upon angiographic occlusion and rising cardiac biomarker levels. Because in some cases of ACO, the artery may spontaneously open by the time of the angiogram, the investigators will need to have surrogate endpoints: this will be culprit lesion OR acute occlusion on the angiogram AND a sufficiently elevated peak troponin, i.e., peak troponin I > 1.0 ng/mL with a 20% change within first 24 hours OR peak troponin T > 5.0 ng/mL, which have been shown to be highly correlated with ACO OR cardiac arrest in a clinical scenario compatible with ACO before blood could be withdrawn for troponin essay.

The sensitivity, specificity and diagnostic accuracy of all these predefined ECG criteria will be sought. Also, sensitivity, specificity and diagnostic accuracy of current established STEMI criteria will be defined. Both short- and long-term mortality of the patients with a diagnosis of STEMI with ACO, STEMI without ACO, NSTEMI with ACO, NSTEMI without ACO and chest pain without acute coronary syndrome will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Admission to emergency department with a clinical picture suggestive of acute coronary syndrome

Exclusion Criteria:

* Absence of documented ECG
* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Siyami Ersek Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aslanger EK, Yildirimturk O, Simsek B, Bozbeyoglu E, Simsek MA, Yucel Karabay C, Smith SW, Degertekin M. DIagnostic accuracy oF electrocardiogram for acute coronary OCClUsion resuLTing in myocardial infarction (DIFOCCULT Study). Int J Cardiol Heart Vasc. 2020 Jul 30;30:100603. doi: 10.1016/j.ijcha.2020.100603. eCollection 2020 Oct. PMID 32775606

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | STEMI | NSTEMI | Normal
Started | 1000 | 1000 | 1000
Completed | 986 | 973 | 1000
Not Completed | 14 | 27 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | STEMI | NSTEMI | Normal | Total
Number analyzed (Participants) | 1000 | 1000 | 1000 | 3000
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (13) | 61 (13) | 48 (16) | 56 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 243 | 334 | 354 | 931
  Male | 757 | 666 | 646 | 2069
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1000 | 1000 | 1000 | 3000
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 1000 | 1000 | 1000 | 3000
Hypertension [Count of Participants; unit: Participants] | 481 | 574 | 195 | 1250
Dyslipidemia [Count of Participants; unit: Participants] | 276 | 367 | 207 | 850
Diabetes [Count of Participants; unit: Participants] | 292 | 371 | 83 | 746
Smoking [Count of Participants; unit: Participants] | 514 | 415 | 483 | 1412
Prior myocardial infarction [Count of Participants; unit: Participants] | 185 | 274 | 89 | 548
Prior percutaneous coronary intervention (PCI) [Count of Participants; unit: Participants] | 150 | 213 | 111 | 474
Prior coronary artery by-pass operation [Count of Participants; unit: Participants] | 55 | 96 | 63 | 214
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 136 (33) | 146 (28) | 139 (24) | 140 (30)
Heart rate [Median (Inter-Quartile Range); unit: bpm] | 80 [53 to 107] | 81 [55 to 107] | 77 [58 to 96] | 79 [69 to 93]
Electrocardiogram to percutaneous coronary intervention time [Median (Inter-Quartile Range); unit: minutes] | 40 [0 to 82] | 2160 [0 to 7230] | NA [NA to NA] — PCI not undertaken in this group | 90 [33 to 2460]
Grace risk score [Median (Inter-Quartile Range); unit: units on a scale] — GRACE risk score is a well known total score system with >140 being high risk. The range for GRACE risk score is from 0 to 263.
  units on a scale | 147 [105 to 189] | 142 [103 to 181] | 129 [85 to 173] | 143 [125 to 166]
Creatinine [Mean (Inter-Quartile Range); unit: mg/dL] | 0.8 [0.5 to 1.1] | 0.9 [0.5 to 1.3] | 0.8 [0.6 to 1.0] | 0.8 [0.7 to 1.0]
Hemoglobin [Mean (Inter-Quartile Range); unit: g/dL] | 13.7 [11.2 to 16.2] | 13.3 [10.6 to 16] | 13.9 [11.4 to 16.4] | 13.6 [12.2 to 14.8]
Admission troponin [Median (Inter-Quartile Range); unit: ng/ml] | 3.462 [0 to 23.017] | 0.403 [0 to 2.276] | 0.002 [0 to 0.005] | 0.155 [0.003 to 2.543]

OUTCOME MEASURES:

1. Primary Outcome: The Sensitivity and Specificity of ECG for Acute Coronary Occlusion.
Description: Determine the sensitivity and specificity of different ECG findings for acute coronary occlusion. The Number of Participants with Type 1a and 1b ECGs, as defined in the study protocol.
Time Frame: Up to 48 hours
Population: The occurrence of type 1a and 1b ECGs in subgroups
Measure: Count of Participants; unit: Participants
Arm/Group | STEMI | NSTEMI | Normal
Number analyzed (Participants) | 1000 | 1000 | 1000
Participants | 767 | 282 | 16

2. Secondary Outcome: The Sensitivity and Specificity of Current "STEMI" Criteria for Acute Coronary Occlusion.
Description: Determine the accuracy of current "STEMI" ECG criteria (as reported in the 4th universal definition of MI) in diagnosing acute coronary occlusion. Type 1a, 1c and 1d ECGs will be included in this group.
Time Frame: Up to 48 hours
Population: THe occurrence of type 1c and 1d ECGs in subgroups
Measure: Count of Participants; unit: Participants
Arm/Group | STEMI | NSTEMI | Normal
Number analyzed (Participants) | 1000 | 1000 | 1000
Participants | 233 | 0 | 3

3. Secondary Outcome: The Sensitivity and Specificity of ECG Without ST-segment Elevation for Acute Coronary Occlusion
Description: Determine the accuracy of ECG interpretation of acute coronary occlusion without STEMI criteria. Only type 1b ECGs will be included in this group.
Time Frame: Up to 48 hours
Population: The occurrence of type 1b ECGs in subgroups
Measure: Count of Participants; unit: Participants
Arm/Group | STEMI | NSTEMI | Normal
Number analyzed (Participants) | 1000 | 1000 | 1000
Participants | 0 | 41 | 5

4. Secondary Outcome: The Specificity of ECG With STEMI Criteria
Description: Explore the rationale for correct ECG interpretation of false positive STEMI criteria. Only type 1c and 1d ECGs will be included in this group.
Time Frame: Up to 48 hours
Population: The sum of type 1c and 1d ECGs in subgroups
Measure: Count of Participants; unit: Participants
Arm/Group | STEMI | NSTEMI | Normal
Number analyzed (Participants) | 1000 | 1000 | 1000
Participants | 233 | 3 | 70

5. Secondary Outcome: The Sensitivity of ECG With STEMI Criteria
Description: Explore the rationale for correct ECG interpretation of false negative STEMI criteria. The occurrence of type 1c ECGs in subgroups will be compared.
Time Frame: Up to 48 hours
Population: The occurrence of type 1c ECGs in subgroups
Measure: Count of Participants; unit: Participants
Arm/Group | STEMI | NSTEMI | Normal
Number analyzed (Participants) | 1000 | 1000 | 1000
Participants | 123 | 3 | 64

6. Secondary Outcome: The Outcome (Mortality) According to ECG Subclassifications (STEMI/NSTEMI/Control Groups)
Description: Compare the outcomes of the patients who are labeled as STEMI and the patients who are labeled as having NSTEMI but have acute coronary occlusion.
Time Frame: Up to one year
Measure: Count of Participants; unit: Participants
Arm/Group | STEMI | NSTEMI | Normal
Number analyzed (Participants) | 986 | 973 | 1000
Participants | 135 | 60 | 1

ADVERSE EVENTS:
Time Frame: 1.5 years
Description: Survival/mortality
Arm/Group | STEMI | NSTEMI | Normal
All-Cause Mortality (participants affected / at risk) | 135/1000 | 60/1000 | 1/1000
Serious Adverse Events (participants affected / at risk) | 83/1000 | 27/1000 | 0/1000
Other Adverse Events (participants affected / at risk) | 0/1000 | 0/1000 | 0/1000
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STEMI (N=1000) | NSTEMI (N=1000) | Normal (N=1000)
In hospital mortality (Cardiac disorders) | 83 (83) | 27 (27) | 0 (0) — Serious event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-04-23): https://cdn.clinicaltrials.gov/large-docs/68/NCT04022668/Prot_SAP_ICF_000.pdf